CLINICAL TRIAL: NCT03702088
Title: Place of the Hevylite Test in the Evaluation of MRD in Myeloma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nice (Other); Hospices Civils de Lyon (Other); CLB de Lyon (Unknown); Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0234
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Myeloma
Keywords: Minimal residual disease; Multi-parametric flow cytometry; Hevylite®
MeSH Terms: conditions — Neoplasms, Plasma Cell; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study aiming at testing the positive predictive value of the Hevylite blood test in detecting minimal residual disease in myeloma compared to an invasive method requiring bone marrow sample by multi-parametric flow cytometry

DETAILED DESCRIPTION:
Multiple Myeloma is a pathology for which treatments are constantly progressing. These treatments allow more and more patients to reach deeper and deeper responses. Currently, it is possible to detect very low levels of disease : this is called the evaluation of minimal residual disease. Its prognostic value is strong.

Two techniques currently prevail in the evaluation of minimal residual disease: high throughput sequencing (NGS) and multi-parameter flow cytometry. They are included in evaluation criteria defined by the International Myeloma Working Group (IMWG). These techniques have the advantage of being very sensitive, reaching 10-5 (cytometry: 50 events among 5 000 000 cells analysed) to 10-6 (NGS). Nevertheless, they are invasive for the patient (medullary specimen), require technical expertise and are not necessarily available in all hospitals.

The development of blood tests would cope with this constraints.

The Hevylite® assay is a simple, sensitive, automated and inexpensive immunologic technique that allows the accurate quantification of total IgG, Total IgG, Total IgA, Total IgA L, Total IgM, and Total IgM in the blood. Given its characteristics, the Hevylite assay could play a role in the definition of MRD and allow evaluation of residual disease in myeloma.

This study aims to evaluate the positive predictive value of the Hevylite test in the evaluation of residual disease in myeloma in comparison with multiparametric flow cytometry on the bone marrow.

ELIGIBILITY:
Inclusion criteria:

-All patients with myeloma in complete response defines as: Absence of monoclonal component on serum and urine electrophoresis Negative immunofixation on serum and urine Normal ratio of free light chains according to the standard Freelite® method

- Any number of treatment lines received

Exclusion criteria:

- No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for myeloma benefiting from a residual disease evaluation by cytometry according to the current practice.
Sampling Method: Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
positive predictive value of the Hevylite test | 1 day
  positive predictive value of the Hevylite test in the evaluation of residual disease in myeloma in comparison with multiparametric flow cytometry on the bone marrow

SECONDARY OUTCOMES:
Sensitivity the Hevylite test | 1 day
  Sensitivity the Hevylite test in the evaluation of residual disease in myeloma in comparison with multiparametric flow cytometry on the bone marrow
negative predictive value of the Hevylite test | 1 day
  negative predictive value of the Hevylite test in the evaluation of residual disease in myeloma in comparison with multiparametric flow cytometry on the bone marrow
specificity of the Hevylite test | 1 day
  specificity of the Hevylite test in the evaluation of residual disease in myeloma in comparison with multiparametric flow cytometry on the bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: Laure Vincent, Md, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France